CLINICAL TRIAL: NCT06733688
Title: A Study to Evaluate the Pharmacokinetics and Definitive Bioequivalence of Tedizolid Phosphate Single Unit Dose Sachet Powder for Oral Suspension Compared to Tedizolid Phosphate Multiple Dose Bottle Powder for Oral Suspension
Brief Title: A Study to Evaluate Oral Formulations of Tedizolid Phosphate in Healthy Participants (MK-1986-043)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1986-043; MK-1986-043 (Other: MSD)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tedizolid Phosphate Oral Formulation 1 (Reference) (Experimental): Participants receive tedizolid phosphate formulation 1 orally.
  Interventions: Drug: Tedizolid Phosphate Oral Formulation 1 (Reference)
- Tedizolid Phosphate Oral Formulation 2 (Test) (Experimental): Participants receive tedizolid phosphate formulation 2 orally.
  Interventions: Drug: Tedizolid Phosphate Oral Formulation 2 (Test)

INTERVENTIONS:
Drug: Tedizolid Phosphate Oral Formulation 1 (Reference) — Oral administration
  Other Names: MK-1986; TR-701 FA
  Arms: Tedizolid Phosphate Oral Formulation 1 (Reference)
Drug: Tedizolid Phosphate Oral Formulation 2 (Test) — Oral administration
  Other Names: MK-1986; TR-701 FA
  Arms: Tedizolid Phosphate Oral Formulation 2 (Test)

SUMMARY:
The goal of the study is to learn what happens to different oral formulations of tedizolid phosphate (MK-1986) in a healthy person's body over time. Researchers want to know if there is a difference in the absorption and elimination of different oral formulations from the healthy person's body.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18.5 and ≤34 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of clinically significant cancer (malignancy)

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the AUC0-Inf of tedizolid.
Area Under the Concentration-Time Curve from Time 0 to the Last Measurable Concentration (AUC0-t) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the AUC0-t of tedizolid.
Maximum Plasma Concentration (Cmax) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the Cmax of tedizolid.

SECONDARY OUTCOMES:
Time to Maximum Plasma Concentration (Tmax) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the Tmax of tedizolid.
Apparent Terminal Half-Life (t1/2) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the t1/2 of tedizolid.
Apparent Volume of Distribution of Tedizolid After Nonintravenous Administration (Vd/F) | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the Vd/F of tedizolid.
Oral Clearance (CL/F) of Tedizolid | At designated time points (up to 3 days postdose)
  Blood samples will be collected to determine the CL/F of tedizolid.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 2 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 2 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com